CLINICAL TRIAL: NCT05617976
Title: Nalbuphine as an Adjuvant to Levobupivacaine in Caudal Analgesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MS 120/2020
Record Dates: First submitted 2022-02-23; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Caudal Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (levobupivacaine only group) (Active Comparator): Caudal block was done in this group using levobupivacaine 0.25% with the dose of 1 ml /kg plus one ml normal saline after induction of general anesthesia.
  Interventions: Procedure: caudal block
- Group L+N(levobupivacaine plus nalbuphen group) (Active Comparator): Caudal block was done in this group using levobupivacaine 0.25% with the dose of 1 ml /kg and nalbuphine 0.1 mg /kg in one ml normal saline after induction of general anesthesia.
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: caudal block — caudal block

SUMMARY:
Caudal anesthesia is the single most important pediatric regional anesthetic technique and is increasingly performed in pediatric regional anesthesia practices. It is preferred in order to relieve intra-operative and postoperative pain in children of all age groups undergoing pelvi-abdominal or lower limbs surgeries using levobupivacaine 0.25%.Various adjuvants have been added to levobupivacaine to prolong postoperative caudal analgesia. Nalbuphine as many opioids can be added in caudal analgesia. This prospective randomized double blind study was done to compare the effects of plain levobupivacaine versus Levobupivacaine plus nalbuphine single-shot for postoperative pain relief in children undergoing hypospadius repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II.
* Age 1-3 years.
* Patients scheduled for hypospadias repair surgeries.

Exclusion Criteria:

* ASA III, IV.
* Signs of infection at site of injection.
* Known coagulopathy disorder.
* Mental and / or developmental retardation.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Quality of Postoperative analgesia | 24 hours
  Face legs activity cry consolablity score (FLACC) (0-10) Score: 0, no pain; 1-3, mild pain; 4-7, moderate pain; 8-10, severe pain
duration of analgesia | 24hours
  Time to first analgesia request (TFAR)

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  total dose of rescue analgesic

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt